CLINICAL TRIAL: NCT01688934
Title: A Phase 2, Randomized, Double-blind, Placebo- and Active-controlled, Parallel-group, Multicenter Study Evaluating the Analgesic Efficacy and Safety of V116517 in Subjects With Moderate to Severe Chronic Pain Due to Osteoarthritis of the Knee
Brief Title: Analgesic Efficacy and Safety of V116517 in Subjects With Moderate to Severe Chronic Pain Due to Osteoarthritis (OA) of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VND2001
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Osteoarthritis, Knee; Pain
Keywords: Pain; Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis | interventions — 4-(3-chloro-5-(1,2-dihydroxyethyl)-2-pyridyl)-N-(5-(trifluoromethyl)-2-pyridyl)-3,6-dihydro-2H-pyridine-1-carboxamide; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- V116517 - 50 mg (Experimental): V116517 50-mg tablets
  Interventions: Drug: V116517 50-mg tablets; Drug: Placebo
- V116517 - 30 mg (Experimental): V116517 30-mg tablets
  Interventions: Drug: V116517 30-mg tablets; Drug: Placebo
- Naproxen 500 mg (Active Comparator): Naproxen 500-mg capsules
  Interventions: Drug: Naproxen 500-mg capsules; Drug: Placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: V116517 50-mg tablets — Taken orally twice daily
  Arms: V116517 - 50 mg
Drug: V116517 30-mg tablets — Taken orally twice daily
  Arms: V116517 - 30 mg
Drug: Naproxen 500-mg capsules — Taken orally twice daily
  Arms: Naproxen 500 mg
Drug: Placebo — Tablets to match V116517 and/or placebo capsules to match naproxen taken orally twice daily

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy of 2 dose levels of V116517 versus placebo.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects with moderate pain due to OA of the knee as their primary pain condition.
2. Subjects with diagnostic criteria for primary pain condition (American college of Rheumatology [ACR] clinical and radiographic criteria):

   * At least 1 of the following in addition to knee pain: age >50, stiffness <30 min, crepitus on active motion, and
   * Kellgren-Lawrence (K-L) grade ≥ 2 radiographic evidence within the past 2 years.

Key Exclusion Criteria:

1. Subjects with chronic pain conditions other than OA of the knee as their predominant pain condition, including gout, pseudo gout, psoriatic arthritis, active Lyme disease, rheumatoid arthritis or any other inflammatory arthritis, fibromyalgia, neuropathic pain conditions, bursitis, or acute injury or signs of active infection in the target pain area.
2. Subjects who cannot or will not agree to stop all concomitant analgesic medications, apart from specified protocol supplemental analgesic medications.
3. Subjects with history of seizures within the past 5 years.
4. Subjects who use opioids more than 4 days per week.
5. Pain-condition-specific exclusions:

   * Subjects who received local pain-control procedures, including intra- articular steroid injection in the study knee or intramuscular steroid injection at any site within 6 weeks of entering the study or hyaluronate injection in the study knee within 12 weeks of entering the study.
6. Subjects who have had arthroscopy on either knee or hip within 6 months of entering the study, or open surgery on either knee or hip within 12 months of entering the study.
7. Active-comparator-related exclusions:

   * Subjects who are allergic to or cannot tolerate naproxen or acetaminophen, including history of NSAID-induced asthma, or nasal polyps;
   * Subjects with history of bleeding disorders or history of documented gastrointestinal ulcer disease.

Other protocol specific inclusion/exclusion criteria may apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster OA Index (WOMAC) Pain Score | Week 4

SECONDARY OUTCOMES:
WOMAC Physical Function Score | Week 4
WOMAC Stiffness Score | Week 4
Modified Brief Pain Inventory - Short Form (mBPI-SF) Severity of Pain and Interference of Pain | Week 4
Patient Global Impression of Change (PGIC) | Week 4
Supplemental Analgesic Medication Use | Over 4 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Compass Research, LLC, Orlando, Florida
  - Compass Research East, LLC, Oviedo, Florida
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - Analgesic Solutions, Natick, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - PMG Research of Charlotte, LLC., Charlotte, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - LION Research, Norman, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLP, Wyomissing, Pennsylvania
  - PMG Research of Bristol, Bristol, Tennessee